CLINICAL TRIAL: NCT05409521
Title: Immediate Effects of Kinesio Taping Applied to the Thoracic Region in Adult Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022/06/02
Record Dates: First submitted 2022-06-02; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Kinesio Taping; Healthy Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tape Group (Experimental): Kinesio taping will be applied on thoracic region
  Interventions: Other: Kinesio taping
- Placebo Group (Placebo Comparator): Placebo taping will be applied on arm region
  Interventions: Other: Placebo taping

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping with the mechanical correction technique will be applied on the thoracic region
  Arms: Tape Group
Other: Placebo taping — Placebo taping with no tension and technique will be applied on the arm
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to search immediate effects of kinesio taping applied to the thoracic region on proprioception, posture and trunk muscle endurance in adult individuals.

DETAILED DESCRIPTION:
Kinesio tape applications are one of the frequently used interventions within the scope of physiotherapy and rehabilitation. Kinesio taping is a non-invasive treatment method performed for several reasons such as reducing pain, relieving abnormal muscle and fascia tension and correcting biomechanical alignment. Kinesio taping consists of muscle, fascia, ligament, mechanic, functional and lymphatic correction techniques depending on therapeutic purposes.

Although kinesio tape applications on different regions such as abdomen or neck may have positive effects on posture, proprioception and trunk muscle endurance, there has not been found any study searching the effectiveness of kinesio taping applied to thoracal region on posture, proprioception and trunk muscle endurance in adult individuals. Thus, there is a need to investigate this issue.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years,
* Volunteer to paticipate to the study

Exclusion Criteria:

* Musculoskeletal pain problems in the last 6 months
* Spinal fractures
* History related to spinal surgery
* Spinal deformity (scoliosis etc)
* Any chronic disease (cancer, diabetes mellitus, hypertension etc. )
* Body mass index>35 kg/m2
* Mental or psychologic problems
* Any dermatologic disease
* Allergy to kinesio tape

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Trunk position sense | immediately after the intervention
  Inclinometer will be positioned at spinous process of 4th thoracic vertebrae during trunk position sense assessment. Subject will be retreated to neutral position and asked to come back taught position while eyes closed. Test will be repeated 3 times and angle of deviation from 30 degree flexion position will be recorded and the average of the results will be taken.

SECONDARY OUTCOMES:
Joint position sense of cervical spine | immediately after the intervention
  Whereas one side of inclinometer positioned at apex of head, other side will be positioned at spinous process of 7th cervical vertebrae during assessment of cervical spine joint position sense. Subject' head will be brought to 300 flexion from neutral position and will be wanted to learn this position. Subject will be retreated to neutral position and asked to come back taught position while eyes closed. Test will be repeated 3 times and angle of deviation from 300 flexion position will be recorded to subject assessment sheet each repetition and average of the results will be taken.
Thoracic kyphosis | immediately after the intervention
  The assessment of thoracic kyphosis will be done using dual digital inclinometer. In order to evaluate thoracic kyphosis, the angle between first thoracic vertebrae and 12th thoracic vertebrae will be measured. As the angle increases, the degree of kyphosis increases.
Head-neck posture | immediately after the intervention
  Head-neck posture will be evaluated with the measurement of cranio- vertebral angle. The angle between 7th cervical vertebrae and tragus will be measured with goniometer to determine cranio- vertebral angle. As the angle decreases, the forward tilt of the head increases.
Trunk extensor muscle endurance | immediately after the intervention
  Trunk extensor muscle endurance will be evaluated with Biering- Sorensen test.Subjects will be asked to lie down on a bed in prone position while trunk positioned outside of the bed until SIAS (spina illiaca anterior superior) level. Lower extremity will be stabilised by researchers. Initially subjects will be asked to extend their trunk to horizontal position (bed level) and then cross their arms on the chest and hold at this position as long as they would. The duration that subjects stayed at the horizontal position without any movement will be calculated with chronometer and recorded as second.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University